CLINICAL TRIAL: NCT01570920
Title: Effects of Regular Brisk Walking in Chronic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2008/04JUIL/193
Record Dates: First submitted 2010-03-30; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Stroke
Keywords: Activity limitations; restriction of participation; chronic stroke survival; physical activity; walking
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- walking (Experimental): a cohort of stroke patients trained during 3 month, based on walking
  Interventions: Behavioral: physical training

INTERVENTIONS:
Behavioral: physical training — walking many times a week

SUMMARY:
Chronic stroke patients (>6 months) fulfilling including criteria were trained during 3 months. The physical training program was based on walking.

DETAILED DESCRIPTION:
Participants had been evaluated 4 times during a long follow-up period of 7 months. Activity limitations were assessed at baseline (enrollment time point), 1 month, 4 months and 7 months later.

ELIGIBILITY:
Inclusion Criteria:

* Stroke onset > or = 6 months
* Able to walk without human assistance (may use walking aid)
* Sign informed consent form
* Approval from physician for participation in study
* Live in Belgium or in Benin

Exclusion Criteria:

* cardiac history of active unstable angina, recent (less than 3 months) myocardial infarction, or congestive heart failure
* orthopedic, circulatory, or chronic pain conditions restricting exercise;
* dementia;
* severe receptive or global aphasia with inability to follow 2-step commands;
* co-morbid non-stroke neurological disorder that impairs mobility (e.g. MS or Parkinson's);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
ACTIVLIM-Stroke (Activity limitations measures) | 7 months
  mainly self-reported outcomes measures

SECONDARY OUTCOMES:
Stroke Impairment | 7 months
  Stroke related impairment are assessed with specific outcomes measures (SIAS, BBS, ...).
Walking ability | 7 months
  Walking ability is assessed throuht walking speed and walking endurance

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Thonnard, PhD, Principal Investigator — Université Catholique de Louvain, Belgium
Locations (1):
- Institut of Neuroscience (IoNS) / UCL, 5375, Brussels, Brussels Capital, Belgium

REFERENCES:
- [Derived] Batcho CS, Stoquart G, Thonnard JL. Brisk walking can promote functional recovery in chronic stroke patients. J Rehabil Med. 2013 Sep;45(9):854-9. doi: 10.2340/16501977-1211. PMID 23974944